CLINICAL TRIAL: NCT01753674
Title: The Effects of the Telomerase Activator TA-65 on Insulin Resistance, Inflammation, and Metabolic Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: non-compliance issues
Sponsor: University of Connecticut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H12-256; TAS-12-035 (Other Grant/Funding Number: TA Sciences Inc)
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Metabolic Syndrome; Insulin Resistance
Keywords: metabolic syndrome, insulin resistance, HDL cholesterol,
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TA-65 (Experimental): TA-65 will be provided to volunteers for 12 weeks, two pills per day of 8 mg each
  Interventions: Dietary Supplement: TA-65
- Placebo (Placebo Comparator): Placebo will be provided to volunteers for 12 weeks, 2 pills per day of 8 mg each.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: TA-65 — TA-65 will be provided to volunteers, 2 pills per day of 8 mg each
  Arms: TA-65
Dietary Supplement: Placebo — Placebo supplement will be provided to volunteers, 2 pills per day of 8 mg each
  Arms: Placebo

SUMMARY:
Our hypothesis is that TA-65, a dietary supplement will help to reduce insulin resistance and plasma glucose in individuals classified with metabolic syndrome.

DETAILED DESCRIPTION:
This is double blind cross over randomized clinical trial. The supplement and placebo will be provided by TA Science, Inc. and prepared as described below. Subjects will be randomly allocated to consume either a daily serving of TA-65 (two capsules per day of 8 mg each) (please see attached label) or a placebo for 12 weeks. Randomization will be done in a sequential manner; the first subject will be allocated to supplement A and the next one to supplement B and so on. After a 3-week washout, they will be allocated to the alternate treatment for additional 12 weeks. Supplements (TA-65 or placebo) will be taken twice daily with a meal.

Participants will be advised not to change their diet or exercise protocols during the 27 week intervention. Volunteers will be required to provide a 5-day dietary record before starting the study, at the end of each supplement period (TA-65 or placebo) and at the end of the washout period. Subjects will have to fill an exercise questionnaire during the same times to ensure that there are no changes in physical activity. Participants will be asked to report to the department every 4 weeks for checking compliance on supplement intake and to assess weight and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria are:

men and women (40-70 y) with metabolic syndrome which means having at least 3 of the following characteristics:

* Blood pressure > 130/85 mm Hg
* plasma glucose > 100 mg/dL
* plasma triglycerides > 150 mg/dL
* HDL cholesterol < 40 mg/dL (men) and < 50 mg/dL (women)
* waist circumference >102 cm (men) and ≥ 88 cm (women)
* Women of childbearing age should be using contraception

Exclusion Criteria:

Exclusion criteria will be

* self-reported diabetes mellitus
* coronary heart disease
* triglycerides greater than 400 mg/dL
* Fasting glucose greater than 126 mg/dL
* Blood pressure greater than 140/100 mmg Hg
* history of stroke
* Use of alcohol at an elevated rate (more than two drinks per day)
* Renal problems
* liver disease
* cancer
* pregnancy and lactation
* severe infectious diseases
* autoimmune disease currently under treatment
* current hormone therapy
* previous treatment with TA-65.
* Intake of glucose-lowering prescriptions
* Use of immunosuppressants, lithium or supplements such as Sulphonylureas (Glucotrol, Amaryl), Thiazolidinedione (Avandia, ACTOS,), Meglitinides (Prandin, Starlix), Biguanides (Metformin), Alpha-glucosidase inhibitors (Precose, Glyset), dipeptidyl peptidase (DPP)-4 inhibitors (Januvia, Onglyza)
* high dose chromium or cinnamon supplements
* Consistent intake of vitamin, mineral, or multivitamin supplements prior to recruitment may be admitted into the study if they plan on maintaining their current supplement program.

However, subjects may not participate if they begin taking a new supplement during the 27-wk study period.

-Subjects will also be asked to refrain from taking any additional supplements, including fish oil, herb and concentrated antioxidant sources.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Plasma insulin levels | 27 weeks
  The supplement is anticipated to decrease insulin resistance in individuals with metabolic syndrome. The investigators will measure plasma insulin and plasma glucose as outcomes measures

SECONDARY OUTCOMES:
plasma HDL cholesterol | 27 weeks
  It is expected that the TA-65 supplement will increase plasma HDL, another characteristic of metabolic syndrome

OTHER OUTCOMES:
blood pressure | 27 weeks
  It is expected that the supplement will decrease blood pressure, another outcome of metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Luz Fernandez, Ph.D., Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Background] Maubaret CG, Salpea KD, Jain A, Cooper JA, Hamsten A, Sanders J, Montgomery H, Neil A, Nair D, Humphries SE; HIFMECH consortium, Simon Broome Research Group. Telomeres are shorter in myocardial infarction patients compared to healthy subjects: correlation with environmental risk factors. J Mol Med (Berl). 2010 Aug;88(8):785-94. doi: 10.1007/s00109-010-0624-3. Epub 2010 Apr 11. PMID 20383691
- See also: Sponsor Company — http://www.tasciences.com/